CLINICAL TRIAL: NCT06956248
Title: Innovating Access to Novel Therapies Through Standardized Prospective Integration of Response Evaluations (IMPACT-INSPIRE)
Acronym: IMPACT-INSPIRE
Status: Recruiting | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: SingHealth Duke-NUS Academic Medical Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024/3309
Record Dates: First submitted 2025-04-30; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor
Keywords: Advanced Cancers; Solid Tumours; Off-label Cancer Therapies; Non-standard Cancer Therapies; Molecular Tumour Board (MTB); Response Assessment; Real-World Data Collection; Precision Oncology; Translational Research; Patient Reported Outcomes (PROs); Quality of Life (QOL); Treatment Outcomes
MeSH Terms: interventions — Off-Label Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population with histologic or cytologic confirmed advanced solid tumours: Histologic or cytologic confirmed advanced treatment refractory solid tumours with no further suitable standard treatment options.
  Interventions: Other: Off-label or non-standard systemic therapies

INTERVENTIONS:
Other: Off-label or non-standard systemic therapies — Off-label systemic treatments and/or relevant clinical trials recommended by the NCCS Molecular Tumour Board (MTB).

SUMMARY:
This observational study aims to assess the outcomes in patients with advanced treatment refractory cancers with matched molecular/precision therapy as per their molecular profiling results after discussion at molecular tumour board.

1. To standardize response assessment and data collection for patients that are receiving off-label or non-standard therapies based on MTB recommendations.

   - Establish a standardized response assessment process and data collection patients that are receiving off-label or non-standard therapies based on MTB recommendations.
2. To demonstrate that it is feasible to standardize investigations and endpoints in this proof-of-concept study.

   * Through standard safety laboratory investigations (FBC, U/E/Cr, LFT)
   * Through standard radiological imaging at 6-12 weeks with the key endpoint being best response during that imaging window, and disease control rate at 6 months.

Hypothesis: Our proposed IMPACT-INSPIRE study hypothesis is that standardised response assessment and data collection in patients with no available therapies receiving off-label systemic therapies, can provide a novel mechanism to assess oncological outcomes in this unique cohort of patients, generate hypothesis, and provide insights to future biomarker-driven drug development

DETAILED DESCRIPTION:
The patient will be observed clinically after informed consent has been obtained. Patients may require more frequent assessment or additional procedures as clinically necessary or as required by the product label.

* Each participant will have undergone comprehensive molecular profiling with results discussed at NCCS molecular tumour board. Where necessary, orthogonal studies/assays may be performed.
* The molecular profiling results will be provided by the referring physician and primary investigator/co-investigator (PI/Co-I). All cases will be presented in the NCCS Molecular Tumour Board (MTB) where there is an adequate quorum of participating members.
* The MTB will analyse the findings and provide a written report to the treating physician on recommended treatments and/or relevant clinical trials; the treating physician makes all treatment decisions.
* The subsequent treatments and treatment responses will be tracked longitudinally during the term of this study, thus linking molecularly informed treatments to specific patient outcomes.
* Translational tissue and plasma may be additionally collected at various timepoints during the study for correlational translational research

ELIGIBILITY:
Inclusion Criteria:

1. Is equal to or greater than 21 years of age;
2. Histologic or cytologic confirmed advanced solid tumours;
3. Patients who have received and failed all standard anticancer therapy (if available) or are unsuitable for further standard anticancer therapy. Cancers with a poor prognosis or low expected response rate to standard treatment (as judged by the investigator on the basis of available evidence) may be screened with respect to an earlier line of treatment;
4. Ability to understand and the willingness to provide written informed consent.

Exclusion Criteria:

1. Specific contraindications to exposure to the off-label or non-standard therapy (as defined by the product label);
2. Other comorbid conditions that may compromise assessing key outcomes or, in the judgement of the clinician, limit the ability of the patient to comply with the protocol.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologic or cytologic confirmation confirmed of advanced refractory solid tumours with no further suitable treatment options.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2027-03-12 (Estimated)

PRIMARY OUTCOMES:
Best objective response rate at 12 weeks | Up to 12 weeks.
  The percentage of participants with best overall response of complete response (CR) or partial response (PR).
Tumour growth rate inhibition | Up to 12 weeks.
  Duration that patient is on experimental therapy as a fraction of the total duration on last line of therapy.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs), Identified and graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 criteria. | From the initiation of protocol therapy, up to 30 days after last dose of off-label or non-standard therapy.
Quality of life thorough AE evaluation or equivalent instruments such as the EORTC QLQ-C30 questionnaire. | Baseline and after every 2 cycles till end of treatment, up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel SW Tan, BSc(Hons), MBBS, MRCP, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided